CLINICAL TRIAL: NCT02151656
Title: Effects of F17464 in Acute Exacerbation of Schizophrenia
Brief Title: F17464 in Acute Schizophrenia Trial
Acronym: FAST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F17464 GE 2 01; 2013-005451-32 (EudraCT Number)
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Mental disorders; Antipsychotic Drugs
MeSH Terms: conditions — Schizophrenia; Mental Disorders | interventions — dopamine D3 receptor antagonist F17464

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- F17464 (Experimental): Oral administration - During 6 weeks - 4 capsules daily
  Interventions: Drug: F17464
- Placebo (Placebo Comparator): Oral administration - During 6 weeks - 4 capsules daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: F17464
  Arms: F17464
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the potential efficacy of oral F17464 in comparison to placebo over 6 weeks in patients with acute exacerbation of schizophrenia. Study design: double-blind, randomized, placebo-controlled, parallel-groups, fixed-dose design, multicentre study.

ELIGIBILITY:
Inclusion Criteria:

Demographic and other characteristics

* Male or female, 18-64 years of age inclusive
* primary diagnosis of schizophrenia undergoing an acute exacerbation with prominent "active phase" symptoms, as described by the Diagnostic and Statistical Manual of Mental Disorders, 4th edition - Text Revision (DSM IV-TR) using the MINI 6.0 (Mini-International Neuropsychiatric Interview) for schizophrenia and psychotic disorders related to DSM IV-TR
* Well-documented diagnosis of schizophrenia for a minimum of 1 year before the screening visit
* Since the diagnosis of schizophrenia, the average number of hospitalisations should be no higher than 2 per year (the minimum duration of hospitalization should be more than 4 days)
* During the year before Visit 1, maximum 3 acute psychotic episodes that required hospitalization or change of antipsychotic medication or other therapeutic intervention
* Adequate clinical response to well-conducted treatment courses during previous acute episodes. A well conducted treatment course is defined as an antipsychotic treatment with the usual doses for at least 4 weeks

Current acute episode

* Structured Clinical Interview for the Positive And Negative Syndrome Scale (SCI-PANSS) with a PANSS total score ≥ 70 to < 120 (at Visit 1 and 2)
* Rating of at least 4 (moderate) on at least 2 of the following 4 PANSS positive symptoms: delusions, hallucinatory behaviour, conceptual disorganization, suspiciousness/persecution
* Clinical Global Impression of Severity (CGI-S) score ≥ 4 (moderate or severe)
* Antipsychotic initiated for this acute episode and/or ongoing chronic antipsychotic treatment, with a maximum of 2 antipsychotics in total needed to be changed (due to inefficacy or safety reasons)
* Hospitalization and/ or treatment for the current psychotic episode for less than 2 weeks prior to Visit 1
* No significant improvement of PANSS total score between enrolment (Visit 1) and inclusion (Visit 2) corresponding to a score improvement < 20% on positive symptoms subscale

Exclusion Criteria:

Related to the pathology

* Patients in their first acute episode of psychosis
* Current schizophrenic episode with predominant negative symptoms
* Patient " known to be refractory " defined as lack of significant improvement (no significant relief of symptoms, and no period of good function) despite adequate courses with at least 3 different antipsychotics medication cycles of an adequate duration (at least 4 weeks) and at adequate dosage during the previous 5 years;
* Schizoaffective disorder, schizophreniform disorder and other psychotic disorders;
* Bipolar I and II disorder
* Pervasive developmental disorder, mental retardation, delirium, dementia, memory impairment and other cognitive disorders that would compromise a reliable assessment according to the investigator's opinion
* Known or suspected borderline or antisocial personality disorder or other DSM IV axis II disorder of sufficient severity to interfere with participation in this study
* History of tardive dyskinesia or chronic extra-pyramidal symptoms (EPS), serotonin syndrome or neuroleptic malignant syndrome
* Major depressive disorder which requires a pharmacological treatment
* At imminent risk of injuring him/herself or others or causing significant damage to property, as judged by the investigator
* Suicidal risk based on the Columbia-Suicide Severity Rating Scale (C-SSRS)

  * Any suicidal behavior in the past year
  * Suicidal ideation of type 4 or 5 in the past month

Related to treatments

* Structured psychotherapy (e.g. cognitive behavioural therapy) started within 6 weeks before visit 1
* Electroconvulsive therapy within 3 months before Visit 1
* Previous lack of response to electroconvulsive therapy
* Treatment ongoing with a depot neuroleptic (even if less than 1 cycle in duration before Visit 1)
* Patient having previous treatment course with clozapine within the 4 months prior to Visit 1
* Requirement of concomitant treatment with any of the prohibited medications
* History of intolerance or hypersensitivity to other drugs of the same chemical class as F17464 or to rescue medications or any history of severe drug allergy or hypersensitivity

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 158 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change of the Positive and Negative Syndrome Scale (PANSS) total score | Day 43
  Change from baseline to Day 43 of the PANSS total score

CONTACTS AND LOCATIONS:
Overall Officials: Françoise TONNER, MD, Study Director — Pierre Fabre Medicament
Locations (27):
- France (2):
  - Nîmes
  - Sotteville-lès-Rouen
- Hungary (3):
  - Balassagyarmat
  - Budapest
  - Gyula
- Latvia (4):
  - Daugavpils
  - Jelgava
  - Liepāja
  - Strenči
- Romania (10):
  - Arad
  - Bucharest
  - Campulum G Muscel
  - Craiova
  - Galati
  - Iași
  - Sibiu
  - Târgovişte
  - Târgu Mureş
  - Timișoara
- Russia (8):
  - Arkhangelsky District
  - Engel's
  - Kazan'
  - Moscow
  - Orenburg
  - Saratov
  - Tomsk
  - Yekaterinburg